CLINICAL TRIAL: NCT01380847
Title: Early Prediction of Chronic Allograft Nephropathy by Non Invasive Monitoring of Urinary Cell mRNAs
Brief Title: Prediction of Chronic Allograft Nephropathy
Acronym: Prefigur
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Centaure (Other); ROTRF (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI 09045
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplantation; Kidney Disease; Kidney Failure, Chronic
Keywords: Kidney Transplantation; Allograft; Kidney failure; Chronic allograft nephropathy; Monitoring; Urine
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — RNA profiling of urinary cells in kidney transplant recipients
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal allograft nephropathy: To evaluate urine from KTRs during the first year post-transplantation to assess whether mRNA levels of genes involved in EMT/fibrogenesis can diagnose and predict CAN, and identify patients at risk of chronic allograft dysfunction
  Interventions: Genetic: mRNAs encoding genes

INTERVENTIONS:
Genetic: mRNAs encoding genes — investigate whether the levels of 21 mRNAs encoding genes involved in EMT/fibrogenesis and the alloimmune response are a sensitive and specific non-invasive diagnostic test for CAN in renal allografts

SUMMARY:
The investigators have shown that epithelial-to-mesenchymal transition (EMT) markers in early protocol biopsies of the renal allograft predicts the progression of fibrosis during the first year post-transplantation.

The investigators will develop a non-invasive approach for predicting fibrosis as a substitute for the invasive allograft biopsy procedure, by longitudinal assessment of the mRNA expression level of genes implicated in EMT/fibrogenesis and inflammation in urinary cells from kidney transplant recipients during the first year post-transplantation.

DETAILED DESCRIPTION:
mRNA profiling of urinary cells is fast evolving as a non-invasive substitute for invasive biopsy procedures employed for predicting renal allograft outcomes. This technique has been successfully used to develop biomarkers of acute rejection, but has not been evaluated for the diagnosis of allograft fibrosis.

The progressive scarring process of an allograft, called chronic allograft nephropathy (CAN), remains the chief cause of kidney transplant failure. We have shown by immunohistochemistry that epithelial changes suggestive of epithelial-to-mesenchymal transition (EMT) in early protocol biopsies predict the progression of CAN during the first year post-transplantation. Our preliminary results suggest that the urinary cell mRNA profile is altered in kidney transplant recipients (KTRs) with CAN.

The purpose of this study is to evaluate urine from KTRs during the first year post-transplantation to assess whether mRNA levels of genes involved in EMT/fibrogenesis can diagnose and predict CAN, and identify patients at risk of chronic allograft dysfunction.

The scientific underpinnings for our hypotheses are provided by (a) data showing that urinary cell mRNAs predict pathological changes (i.e., acute rejection) in renal allografts; and (b) our previous studies suggesting that CAN is characterized by altered urinary cell mRNA levels.

Our specific aims are to (1) investigate whether the levels of 21 mRNAs encoding genes involved in EMT/fibrogenesis and the alloimmune response are a sensitive and specific non-invasive diagnostic test for CAN in renal allografts; (2) determine whether mRNA profiles of sequential urine specimens can predict the development of CAN during the first year post-transplantation; and (3) determine whether mRNA profiles of sequential urine specimens predict the subsequent development of graft dysfunction as assessed by estimated GFR at 12, 24 and 36 months after transplantation.

Eligible patients will be consecutive KTRs from Necker Hospital during one year (n≈180). Urine samples will be collected at 1, 3, 6, 9 and 12 months post-transplantation, and 21 mRNAs involved in EMT/fibrogenesis and the alloimmune response will be quantified by PCR. Allograft fibrosis will be quantified by image analysis, developed in our unit. Urinary cell mRNA profiles will be correlated with data from protocol biopsies (3 months and 1 year) and glomerular filtration rate (GFR) at 1 and 3 years. Diagnostic and prognostic accuracy of mRNA levels will be determined.

The identification of molecular markers of CAN may allow for early diagnosis of CAN (before the onset of fixed renal injury) and thus the development of specific therapeutic interventions.

ELIGIBILITY:
Inclusion criteria :

* male and female adult recipients
* patients undergoing primary or re-do deceased-donor or living-donor kidney transplantation
* ability to provide informed consent

Exclusion criteria :

* patients undergoing combined organ transplantation
* Contraindication to protocol allograft biopsy
* Inability or unwillingness of a participant to provide informed consent.
* HCV infected
* HIV infected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients from Necker Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04-19 (Actual); Study Completion 2012-04-19 (Actual)

PRIMARY OUTCOMES:
Renal allograft fibrosis | 2 years
  Renal allograft fibrosis at one year posttransplantation

SECONDARY OUTCOMES:
Renal allograft nephropathy | 4 years
  Progression of renal allograft fibrosis between 3 months and one year posttransplantation Renal allograft function at 3 year posttransplantation

CONTACTS AND LOCATIONS:
Overall Officials: Dany Anglicheau, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Hospital, Paris, France

REFERENCES:
- [Result] Galichon P, Amrouche L, Hertig A, Brocheriou I, Rabant M, Xu-Dubois YC, Ouali N, Dahan K, Morin L, Terzi F, Rondeau E, Anglicheau D. Urinary mRNA for the Diagnosis of Renal Allograft Rejection: The Issue of Normalization. Am J Transplant. 2016 Oct;16(10):3033-3040. doi: 10.1111/ajt.13891. Epub 2016 Jul 8. PMID 27232948